CLINICAL TRIAL: NCT05102916
Title: Swiss Registry for Neuromuscular Disorders (Swiss-Reg-NMD)
Brief Title: Swiss Registry for Neuromuscular Disorders
Acronym: Swiss-Reg-NMD
Status: Recruiting | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: University Children's Hospital Basel (Other); Insel Gruppe AG, University Hospital Bern (Other); University of Lausanne Hospitals (Other); Ente Ospedaliero Cantonale, Bellinzona (Other); University Children's Hospital, Zurich (Other); University Hospital, Zürich (Other); SwissPedNet - Swiss Research Network of Clinical Pediatric Hubs (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2018-00289
Record Dates: First submitted 2021-10-20; First posted 2021-11-02 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: SMA; DMD; BMD; IMD; Congenital Muscular Dystrophy
Keywords: DMD; BMD; IMD; SMA; LAMA2; COL-6; CMD; NMD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 80 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient population: Children, adolescents and adults diagnosed with a NMD (DMD/BMD/IMD; SMA; COL-6; LAMA-2) who are treated or living in Switzerland.

SUMMARY:
The Swiss Patient Registry for DMD/BMD and SMA was launched in 2008 in order to give Swiss patients access to new therapies. It was founded with the financial support of several patient organizations and research foundations. Since 2008, children, adolescents and adults with DMD, BMD and SMA are registered with the help of all major muscle centers in Switzerland. After nearly ten years of activity, the Swiss Patient Registry for DMD/BMD and SMA implemented several adaptations in 2018 to meet current and future expectations of patient's organizations, health authorities and research organizations.

DETAILED DESCRIPTION:
Background:

The 'Swiss registry for neuromuscular disorders' (Swiss-Reg-NMD) collects medical information from people with neuromuscular disorders. It is led by specialized physicians from all over Switzerland and located at the Institute of Social and Preventive Medicine (ISPM) in Bern. The registry includes children and adults living or treated in Switzerland who are diagnosed with Duchenne-Becker Muscular Dystrophy (DMD/BMD), Spinal Muscular Atrophy (SMA), merosin-deficient muscular dystrophy also called LAMA2-related muscular dystrophy (MDC1A respectively LAMA2) ) and Collagen 6 related muscular dystrophy.

The Swiss Registry for neuromuscular disorders was initially founded in 2008 to give Swiss patients with a neuromuscular disease access to new therapies. In 2018, the registry was reorganized to meet new legal requirements and expectations of patients and research organizations. The Swiss Ethics Commission approved the project (project ID: 2018-00289, observational study, risk category A).

NMDs are rare diseases with few patients scattered across the country. A national patient registry with a centralized registration facilitates the participation of Swiss patients in therapeutic trials and the creation of Swiss trial sites.

Objectives:

Primary objectives of the Swiss-Reg-NMD project are:

1. Establish a representative population-based Swiss cohort of children, adolescents and adults with NMDs
2. Provide epidemiological data to investigate the incidence, prevalence, spectrum of diagnosis, survival rates and mortality of NMDs in Switzerland
3. Provide a platform for clinical research:

   1. Offer a resource to recruit Swiss patients in current and future national and international therapeutic trials or observational studies
   2. Offer a resource to facilitate the establishment of therapeutic trial sites in Switzerland
   3. Answer questions in the following areas: health, health care, social-, educational-, professional-, economic aspects, and quality of life
   4. Offer a resource for post-marketing surveillance (effects and side effects of therapies/treatments)
4. Provide a platform for communication:

   1. Promote the exchange of knowledge between clinics, researchers, therapists and national and cantonal health authorities in particular regarding standards of care
   2. Facilitate national and international collaborations, in particular with the international registry of TREAT-NMD and the upcoming Swiss Registry for Rare Diseases

Inclusion/exclusion criteria:

All children, adolescents and adults living or treated in Switzerland who are diagnosed with a NMD. The diagnosis needs to be confirmed, whenever possible, by genetic testing, or at least by biopsy and/or electroneuromyography, according to international standards for the diagnosis of the given NMD. Once the diagnosis is established, there is no specific exclusion criteria.

Currently, patients with SMA, DMD/BMD, merosin-deficient muscular dystrophy also called LAMA2-related muscular dystrophy (MDC1A respectively LAMA2) and Collagen 6 related muscular dystrophy are included.

Procedure:

After a NMD diagnosis, the treating physician informs the patient and the parents (if the patient is still a child) during a consultation in a clinic or practice in writing and orally about the Swiss-Reg-NMD. The patient/parents who wish to participate sign the consent form and the patient is registered in the Swiss-Reg-NMD. If the patient/parents do not wish to participate, only a minimal anonymous data set is recorded.

The following data will be collected:

* Medical data
* Data from questionnaires for patients and families
* Data from links to routine statistics and other medical registries

Clinical data (report of new cases and follow-up reports): NMD subtype, severity, and associated conditions; Comorbidities; Medical care and medication; Therapies; (Serious) adverse events; Hospitalisations; Motor Function Assessments; Socio-demographic characteristics.

Questionnaire data: We will collect data through questionnaires with a focus on (but not exclusively):

* Health related questions like nutrition, sleep, pain
* Health behaviours (e.g., physical activity, smoking)
* Medical equipment use (type, usage, satisfaction)
* Treatments and therapies: frequency, intensity, start, types
* Quality of life and participation (involvement in a life situation)
* Social-economic factors
* Education (early childhood education, school, professional integration)
* Patient/caregiver reported outcomes
* Needs and concerns of persons with NMDs and their families

Routine data and linkages: e.g. Federal Statistical Office (e.g. birth registry, cause of death statistics, hospital statistics); Swiss National Cohort (socioeconomic data, family information); other medical registries (e.g. rare disease registry); Communities of residence (vital status, date of death, address).

Funding:

Schweizerische Muskelgesellschaft; ASRIMM, Association Suisse Romande Intervenant contre les Maladies neuromusculaire; MGR, Associazione malattie genetiche rare della svizzera italiana; fsrmm, schweizerische stiftung für die erforschung der muskelkrankheiten; SMA Schweiz; Duchenne Schweiz; Amicus Therapeutics; Avexis; Biogen; ITF Pharma; Novartis; Pfizer, PTC Therapeutics; Roche; Sanofi; Sarepta.

Data protection:

Data generation, transmission, storage and analysis of health related personal data within this project will follow strictly the current Swiss legal requirements for data protection. Data analyses will always be done using pseudonymised datasets. Health related personal data captured during this project are strictly confidential. Project data shall be handled with uttermost discretion and only be accessible to authorized personnel. Direct access to source documents will be permitted for purposes of monitoring, audits or inspections. The data protection concept of ISPM ensures the secure handling of all sensitive data at ISPM and within Swiss-Reg-NMD. The Swiss-Reg-NMD team is responsible for the implementation and compliance with the confidentiality and data security measures.

ELIGIBILITY:
Inclusion Criteria:

* Children, adolescents and adults diagnosed with a NMD
* Who are living or treated for a NMD in Switzerland, and
* Who gave informed consent

Exclusion Criteria:

* None if diagnosis is confirmed, whenever possible, by genetic testing, or at least by biopsy and/or electroneuromyography, according to international standards for the diagnosis of the given NMD.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals living or treated in Switzerland with a diagnosis of a NMD. Currently, Spinal muscular atrophy, Duchenne muscular dystrophy, Merosin negative congenital muscular dystrophy MDC1A and Collagen 6 related muscular dystrophy are included. In the future, patients with other NMDs (e.g. Charcot-Marie-Tooth neuropathy, Myotonic Dystrophy or rare myopathies) may also be included if it appears relevant to clinicians and researchers active in the field of NMDs, patient organisations, and public health representatives.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2071-01-01 (Estimated); Study Completion 2071-01-01 (Estimated)

PRIMARY OUTCOMES:
Personal data | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Registering and updating patients personal data
Initial symptoms | At diagnosis
  Initial symptoms
Age at initial symptoms and diagnosis | At diagnosis
  Age at initial symptoms and diagnosis
Family history | At diagnosis
  Other affected family members
Investigations | At diagnosis
  Type of investigations for diagnosis
Diagnosis | At diagnosis
  Mutation
Change of living status | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Date of death
Change of living status II | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Cause of death
Change in height | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Registering height
Change in weight | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Registering weight
Change in head circumference | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Registering head circumference
Change in motor development and motor functions | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Registering motor development and function (motor function scales)
Change in musculoskeletal system | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Assessing change in musculoskeletal system over time
History of surgeries | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Registering surgeries
Change in cardiac function | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Registering cardiac function
Change in pulmonary function | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Registering pulmonary function
Change in nutritional habits | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Registering feeding habits
Change in cognition | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Assessing mental ability using tests, including language
Change in education | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Registering type of education
Change in therapies | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Registering therapies
Change in orthopaedic situation | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Assessing use of orthopaedic resources
Change in treatments | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Registering treatments
Change in side effects | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Registering side effects of treatments
Change in comorbidities | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Registering comorbidities
History of hospitalizations | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Registering hospitalizations
Change in disease specific markers | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Registering change in disease specific markers
Change in epilepsy | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Registering epilepsy
History of participation in clinical trials and research studies | Baseline medical information, follow-up data collection at regular intervals (at diagnosis, then at least annually, up to 80 years)
  Registering participation in current/past clinical trials and research studies
Questionnaire data | 0-80 years
  Questionnaires focusing on specific research questions (Health-related questions, health behavior, medical equipment, treatments and therapies, quality of life, participation, social-economic factors, academic information, patient/caregiver reported outcomes, needs, concerns)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia E Kuehni, Prof. MD, Principal Investigator — Institute of Social and Preventive Medicine (ISPM), University of Bern
Locations (19):
- Switzerland (19):
  - Cantonal Hospital Aarau, Aarau, Canton of Aargau
  - Pediatric Institute of Southern Switzerland, Ospedale San Giovanni, Bellinzona, Canton Ticino
  - Neuro Centre of Italian Switzerland, Ospedale Regionale di Lugano, Lugano, Canton Ticino
  - University Hospital Lausanne CHUV, Children's Hospital, Lausanne, Vaude
  - University Hospital Lausanne CHUV, Lausanne, Vaude
  - University Children's Hospital Basel, Basel
  - University Hospital Basel, Basel
  - Inselspital Bern, Children's Hospital, Bern
  - Inselspital Bern, Bern
  - Institute of Social and Preventive Medicine (ISPM), University of Bern, Bern
  - University Hospitals of Geneva, Children's Hospital, Geneva
  - University Hospitals of Geneva, Geneva
  - Cantonal Hospital of Lucerne LUKS, Lucerne
  - Cantonal Hospital of Lucerne, LUKS, Lucerne
  - Private Practice Alpenquai, Lucerne
  - Cantonal Hospital of Eastern Switzerland, Sankt Gallen
  - Children's Hospital of Eastern Switzerland, Sankt Gallen
  - University Hospital Zuerich, Children's Hospital, Zurich
  - University Hospital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Researchers who wish to develop a nested study need to submit a proposal to the Swiss-Reg-NMD and request permission. A concept sheet describing the planned analyses must be approved by the Swiss-Reg-NMD Steering Board. Nested studies might need separate ethics permission.

REFERENCES:
- See also: Website of the registry — http://www.swiss-reg-nmd.ch